CLINICAL TRIAL: NCT01388608
Title: Correlation of Standard Disease Activity Parameters in Rheumatoid Arthritis With Activities of Daily Living Measured With the Step Activity Monitor, Based on the Influence of Etanercept Therapy on the Disease Activity
Brief Title: Standard Disease Activity Parameters and Step Activity in Patients With Rheumatoid Arthritis Receiving Etanercept
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: StepcountETN
Record Dates: First submitted 2011-06-28; First posted 2011-07-06 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; etanercept; step activity measure
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients receiving etanercept: Patients with active rheumatoid arthritis (RA) who are eligible to a treatment with etanercept.

SUMMARY:
Data on activities of daily living in patients with rheumatoid arthritis are assessed mainly be the health assessment questionnaire (HAQ). The HAQ generates data by subjective variables. It would be desirable and advantageous to add objective tools reflecting patients' activities to the outcome parameters in rheumatoid arthritis. The StepWatch™ activity monitor (SAM) in an ankle worn step counter and an accurate instrument to measure real world ambulatory activity. The investigators purpose was to investigate whether activities of daily living measured by SAM increase during a therapy with the TNF-alpha inhibitor etanercept in patients with active rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
In the past decade treatment strategies for rheumatoid arthritis (RA) have changed dramatically. Today far more therapeutic options are available. Patients are being treated earlier and more aggressive than in the past.

These processes have had an influence on the outcome of patients with RA and on the way they are being evaluated.

Outcome variables are disease aspects or consequences that develop over the course of RA. The HAQ score has been shown to be a good predictor of patients outcome in RA. However, the HAQ ist a questionnaire and the score is influenced by subjective factors.

The Step Watch Activity monitor (SAM)is a highly accurate accelerometer-based step monitor. The SAM provides a detailed profile of the number of steps taken by a subject. It is a small unobtrusive device which is worn laterally at the right ankle. It weights only 65 grams and uses 2D accelerometry.

The SAM can provide objective information about activities of daily living.

Etanercept is a recombinant fully human TNF-receptor p75-Fc fusion protein. Numerous studies with etanercept have shown the clinical efficacy. This can be demonstrated by various disease activity scores (e.g the DAS28). In addition there is strong evidence that etanercept improves disability measured by the HAQ.

There are only few publications reporting about measuring physical activity in patients with joint diseases; all of these include patients with osteoarthritis.

Our aim is to include patients with active RA who receive etanercept. These patients are asked to wear the SAM for 7 days before treatment and 4 weeks and 12 weeks after initiation of therapy with etanercept. The step activity measured by the SAM will be correlated with the the clinical sore DAS28 and the HAQ.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis (Disease activity score -DAS28 > 3.2) who are eligible to a treatment with etanercept.
* Age 18 and older
* Male or female

Exclusion Criteria:

* Contraindications against a therapy with etanercept
* Patients not able to comply with the requirements of the protocol

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active rheumatoid arthritis, who are eligible to a treatment with etanercept according to the local german guidelines
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the step counts during a therapy with etanercept in patients with active rheumatoid arthritis | at baseline, after 4, and after 12 weeks for
  During the therapy with etanercept steps will be counted by the Step watch monitor (SAM) for 7 days before therapy(baseline), after 4 weeks, and after 12 weeks.

SECONDARY OUTCOMES:
Correlation of the step counts with the health-assessment-questionnaire and the disease activity measured by DAS28 during a therapy with etanercept | Baseline, week 4 and week 12
  The results of the step watch monitor will be correlated to the results of the the health-assessment-questionnaire (HAQ) and DAS28 under the therapy with etanercept.
  We will measure the step activity by SAM at basline, week 4 and week 12 after initiation of etanercept. At the same time we will will measure the health-assessment-questionnaire (HAQ)and the disease activity score (DAS28).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Willeke, MD, Principal Investigator — University Hospital Muenster, Department of Medicine D, Section for rheumatology
Locations (1):
- University Hospital Muenster, Münster, Germany